CLINICAL TRIAL: NCT03717584
Title: A Cohort Study of the Intestinal Microbiota of Premature Infants
Status: Active, not recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 888501; UCD#888501-3 (Other: UC Davis)
Record Dates: First submitted 2018-07-10; First posted 2018-10-24 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Necrotizing Enterocolitis; Bronchopulmonary Dysplasia; Growth Failure
Keywords: microbiota; metabolome; lipidome
MeSH Terms: conditions — Enterocolitis, Necrotizing; Bronchopulmonary Dysplasia; Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Infant blood, urine,saliva, stomach fluid, poop, and mother's milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Premature infants are at risk for a variety of diseases, the investigators would like to learn more about why some premature babies are at higher risk and some are protected from these diseases.

Scientists at UC Davis and other universities have developed new ways to measure the bacteria and a large number of small molecules in specimens of infant blood, urine, stomach fluid and poop and in mother's milk. These discoveries allow us to consider questions that were impossible to answer before these new techniques were developed. One such question is whether the bacteria in the poop of a premature baby can help us predict the baby's risk for developing infection or a common and serious disease of premature infants called necrotizing enterocolitis. A second question is whether the DNA of a premature baby (obtained from saliva with a q-tip) can predict higher risk for diseases of premature babies.

DETAILED DESCRIPTION:
Samples from eligible infants will be collected and stored for future comparisons. These samples include stool specimens from a messy diaper twice weekly, urine samples from cotton balls in the diaper once weekly, a small sample of stomach fluid once a week just prior to a feeding obtained through the feeding tube, a sample of mom's milk once a week, left-over blood from lab draws, and a sample of saliva on one occasion.

The analysis of key specimens from this cohort will allow us to study the impact of the bacteria in the intestines on outcomes like growth and common diseases of premature infants.

ELIGIBILITY:
Inclusion Criteria:

* gestational age < 33 weeks at birth

Exclusion Criteria:

* none

Max Age: 33 Weeks | Sex: All
Age Groups: Child
Study Population: All mothers in preterm labor in the labor and delivery ward for whom a consultation by the neonatology group is requested will be screened for eligibility. All premature infants admitted to the NICU will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-12-23 (Actual); Primary Completion 2027-03-05 (Estimated); Study Completion 2027-03-05 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of necrotizing enterocolitis | up to 20 weeks, from the time of enrollment until the time of discharge from the neonatal intensive care unit (NICU)
  How many infants in the cohort develop stage 2 or stage 3 necrotizing enterocolitis by Bells modified criteria

SECONDARY OUTCOMES:
Diagnosis of bronchopulmonary dysplasia | up to 20 weeks, from the time of enrollment until the time of discharge from the NICU
  How many infants in the cohort develop mild, moderate, or severe bronchopulmonary dysplasia based on the criteria outlined by Jobe in 2001
Diagnosis of growth failure | up to 20 weeks, from the time of enrollment until the time of discharge from the NICU
  How many infants in the cohort demonstrate growth failure as defined by a decrease in weight z score by greater than 1 from day of life 7 to day of discharge. Outcome neutral language does not apply here as we are focusing on those infants with poor growth compared to infants with normal or excessive growth

CONTACTS AND LOCATIONS:
Overall Officials: Mark Underwood, MD, Principal Investigator — UC Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mai V, Young CM, Ukhanova M, Wang X, Sun Y, Casella G, Theriaque D, Li N, Sharma R, Hudak M, Neu J. Fecal microbiota in premature infants prior to necrotizing enterocolitis. PLoS One. 2011;6(6):e20647. doi: 10.1371/journal.pone.0020647. Epub 2011 Jun 6. PMID 21674011
- [Background] Claud EC, Keegan KP, Brulc JM, Lu L, Bartels D, Glass E, Chang EB, Meyer F, Antonopoulos DA. Bacterial community structure and functional contributions to emergence of health or necrotizing enterocolitis in preterm infants. Microbiome. 2013 Jul 10;1(1):20. doi: 10.1186/2049-2618-1-20. PMID 24450928
- [Background] Jobe AH, Bancalari E. Bronchopulmonary dysplasia. Am J Respir Crit Care Med. 2001 Jun;163(7):1723-9. doi: 10.1164/ajrccm.163.7.2011060. No abstract available. PMID 11401896
- [Derived] Larke JA, Kuhn-Riordon K, Taft DH, Sohn K, Iqbal S, Underwood MA, Mills DA, Slupsky CM. Preterm Infant Fecal Microbiota and Metabolite Profiles Are Modulated in a Probiotic Specific Manner. J Pediatr Gastroenterol Nutr. 2022 Oct 1;75(4):535-542. doi: 10.1097/MPG.0000000000003570. Epub 2022 Jul 25. PMID 35881967
- See also: Learn more or sign up for the study here! — https://studypages.com/s/learning-more-about-premature-infants-803902/